CLINICAL TRIAL: NCT05646082
Title: Preliminary Assessment of Safety and Tolerability of Dostarlimab in Combination Antiretroviral Therapy (cART) Refractory HIV Associated Kaposi Sarcoma
Acronym: STARKAP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21IC6896
Record Dates: First submitted 2022-11-22; First posted 2022-12-12 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Refractory HIV Associated Kaposi Sarcoma
MeSH Terms: interventions — dostarlimab; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: Dostarlimab in Combination Antiretroviral Therapy

INTERVENTIONS:
Drug: Dostarlimab in Combination Antiretroviral Therapy — Patients will receive dostarlimab at the fixed dose of 500 mg dose Q3W for the first 4 doses followed by a fixed 1000 mg dose Q6W until week 48 of treatment.

SUMMARY:
This is a phase 1b, open label, single arm study evaluating the safety and tolerability of the drug dostarlimab in combination antiretroviral therapy (cART) refractory HIV-associated Kaposi Sarcoma (KS), a rare type of cancer usually seen in people with the HIV infection.

Dostarlimab is a type of immunotherapy, and is a monoclonal antibody that has been designed to inhibit the receptor programmed death-1 (PD-1). One of the two ligands for PD-1 has been shown to be upregulated in KS patients, the PDL-1 ligand. By preventing PDL-1 form binding to PD-1, dostarlimab increases the body's immune response to attack more cancer cells.

The safety profile of dostarlimab in this specific cancer has not been explored. The primary aim of this study is therefore to provide confirmatory evidence of safety of dostarlimab in KS patients and to preliminary evaluate its effects on HIV reservoirs and assess how it causes its anti-cancer effects through studying tumour tissue before and after treatment.

This study will be conducted in two parts and will recruit a total of up to 20 patients.

Upon completion of screening investigations inclusive of a fresh tumour biopsy within a 28-days window, patients will receive dostarlimab at the fixed dose of 500 mg dose every 3 weeks for the first 4 doses followed by a fixed 1000 mg dose every 6 weeks. Treatment will be continued until loss of clinical benefit, unacceptable toxicity, patients' withdrawal or completion of a total of 48 weeks of treatment. Part 1 will consist of 6 patients being dosed and observed for toxicity for 21 days following first dose. A trial steering committee will evaluate any treatment related adverse events (AEs) and dose-limiting toxicities (DLTs) reported before deciding on whether to continue onto part 2, where a further 14 patients may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of Kaposi Sarcoma.
2. Available pretreatment biopsy, either fresh (optimal) or archival (acceptable).
3. Established on cART for at least 3 months and no symptomatic or laboratory AE associated with cART > grade 1 by CTCAE criteria v 5.0.

   Note: modifications of cART during screening are allowed provided patients meet all other eligibility criteria and are on effective new regimen for at least 2 weeks.
4. Have an HIV VL<200 cp/ml and CD4+ T-cell count >100/mm3 at screening.
5. Have disease that is measurable by modified AIDS Clinical Trial Group (ATCG) Kaposi sarcoma response criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
7. Be of ≥ 18 years of age
8. Have adequate haematological and organ function, defined as follows:

   Absolute neutrophil count >1.500/mcL, Platelet count >100.000/mcL, Haemoglobin >90 g/L, Total bilirubin ≤1.5x upper limit of normal (ULN) or ≤2xULN for patients with Gilbert's syndrome or on HIV protease inhibitors, Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤2.5x ULN (up to 5x ULN if liver metastases are present), Serum creatinine ≤2.5x ULN or creatinine clearance (CrCl) >60 ml/min in subjects with serum creatinine ≤1.5x ULN. Calculation of CrCl should follow institutional standards.

   International normalized ratio (INR) or prothrombin time (PT) ≤1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) ≤1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
9. Female participants must have a negative serum pregnancy test within 72 hours prior to taking study treatment if of childbearing potential and agree use a highly effective method of contraception from screening through 120 days after the last dose of study treatment or is of nonchildbearing potential. Nonchildbearing potential is defined as follows (by other than medical reasons):

   * ≥45 years of age and has not had menses for >1 year
   * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
   * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use an adequate birth control method throughout the study, starting with the screening visit through 120 days after the last dose of study treatment. See Section 5.4 for a list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
10. Participant must agree to not breastfeed during the study or for 90 days after the last dose of study treatment.
11. Male participant agrees to use a highly effective method of contraception (see Section 5.4 for a list of acceptable birth control methods) starting with the first dose of study treatment through 120 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
12. Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

1. Participant is simultaneously enrolled in any interventional clinical trial.
2. Participant has received anti-cancer therapy (chemotherapy, radiation therapy, immunotherapy or biologic therapy) including investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy. There should be no evidence of treatment-related adverse events > grade 1 by CTCAE criteria.
3. Major surgery within 3 weeks prior to initiating protocol therapy. Study participant must have recovered from any adverse events relating to surgery.
4. Known active tuberculosis (TB) in the first 6 weeks of treatment.
5. Known active Immune Reconstitution Inflammatory Syndrome (IRIS) related to opportunistic pathogens.

   Note: Patients with previous history of IRIS that has fully resolved at the time of screening are eligible.
6. Known history of active uncontrolled hepatitis C virus (HCV) infection, defined as detectable plasma HCV RNA.

   Note: patients with positive HCV serology but negative HCV RNA or those successfully treated for HCV are eligible.
7. Known history of active uncontrolled hepatitis B virus (HBV) infection, defined as detectable plasma HBV DNA in absence of therapy.

   Note: patients with HBV serology indicating immunization (i.e. positive hepatitis B surface antibody, HBsAb and negative core antibody HBcAb), patients with fully resolved acute HBV infection and those with chronic HBV infection adequately treated with antiviral therapy are eligible.
8. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan.
10. Prior therapy with anti-PD-1/PD-L1 and/or anti-CTLA-4 therapy either alone or in combination with other agents.
11. Receipt of live vaccines within 30 days before the first dose of trial treatment and while participating in the trial; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, seasonal flu, H1N1 flu, rabies, bacillus Calmette-Guerin (BCG), and typhoid vaccine.
12. Known hypersensitivity to dostarlimab components or excipients.
13. Evidence of serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection.
14. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Principal Investigator (PI).
15. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
17. Participant has leptomeningeal disease, carcinomatous meningitis, symptomatic brain metastases, or radiologic signs of CNS hemorrhage.

    Note: Participants with asymptomatic brain metastases (i.e, off corticosteroids and anticonvulsants for at least 7 days) are permitted.
18. Systemic steroid therapy or any other form of immunosuppressive therapy that cannot be discontinued within 7 days prior to initiating protocol therapy.

    Note: inhaled, topical corticosteroid and replacement corticosteroid therapy at physiological doses is permitted.
19. Participant has a history of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | 90 days after treatment
  The safety and tolerability of pembrolizumab will be assessed by recording the incidence of adverse events (AEs) using National Cancer Institute Common Terminology Criteria for Adverse Events NCI CTC criteria v.5.0

SECONDARY OUTCOMES:
Improvement of progression-free survival rate (efficacy) | week 13, 31 and end of treatment
  The Objective Response rate (ORR) evaluated by modified AIDS Clinical Trial Group (ACTG) Kaposi sarcoma (KS) response criteria and by Response Evaluation Criteria In Solid Tumours (RECIST) v1.1 For patients with visceral involvement

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea & Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided